CLINICAL TRIAL: NCT00992628
Title: Measurement of Forces Applied Using a Macintosh Direct Laryngoscope Compared to GlideScope Video Laryngoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Richard Cooper MD, Principal Investigator, Toronto General Hospital, University Health Network
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UHN REB 09-0262-B
Record Dates: First submitted 2009-05-01; First posted 2009-10-09 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2011-04

CONDITIONS: Endotracheal Intubation; Laryngoscopy
Keywords: GlideScope Video Laryngoscope; Macintosh Direct Laryngoscope; Intubation; Applied Forces; Elective surgery where endotracheal intubation required
MeSH Terms: interventions — Laryngoscopes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Macintosh (direct vision) laryngoscope (Active Comparator): Macintosh (direct vision) laryngoscope
  Interventions: Device: Macintosh (direct vision) laryngoscope
- GlideScope videolaryngoscope (indirect vision) (Active Comparator): GlideScope videolaryngoscope (indirect vision)
  Interventions: Device: GlideScope videolaryngoscope (indirect vision)

INTERVENTIONS:
Device: Macintosh (direct vision) laryngoscope — Macintosh (direct vision) laryngoscope
  Arms: Macintosh (direct vision) laryngoscope
Device: GlideScope videolaryngoscope (indirect vision) — GlideScope videolaryngoscope (indirect vision)
  Arms: GlideScope videolaryngoscope (indirect vision)

SUMMARY:
Patients undergoing surgery or intensive care management often require a tube to be inserted into the trachea allowing lung ventilation. Usually a laryngoscope is used to allow visualisation of the larynx and facilitate intubation.

During direct laryngoscopy, the blade of the laryngoscope is inserted into the patient's mouth and the structures pulled upwards out of the line of vision. If visualisation is difficult, users often exert excess force on the tissues to obtain an adequate view. Generally the applied force is evaluated by the patient's stress response such as increased heart rate, blood pressure or plasma cortisol levels. These changes, while important, may be confounded by a variety of patient factors, as well as anaesthesia. An increased force may also be associated with tissue trauma, dental damage, and prolonged attempts.

The investigators' objective is to compare the force exerted on patient's tissues by the Macintosh laryngoscope and GlideScope video-laryngoscope. Video-laryngoscopes may be associated with the application of reduced force to the soft tissues of patients during intubation. While this is a common contention, it has not been proven. The GlideScope has a micro camera in the distal portion of the blade meaning a direct line of vision is not required. An adequate view can therefore be obtained with less displacement of tongue tissue. If the force exerted by the video laryngoscope is less, this would have beneficial implications by reducing stress response, neck movement, and trauma.

ELIGIBILITY:
Inclusion Criteria:

* age > 18years
* ASA 1-2
* elective surgery
* endotracheal intubation required (with non-depolarising muscle relaxant)
* signed informed consent

Exclusion Criteria:

* lack of informed consent
* endotracheal intubation not required
* ASA 3-5
* symptomatic gastro-oesophageal reflux
* rapid sequence intubation
* other method of intubation indicated eg fibreoptic, awake tracheostomy
* cervical spine instability
* unstable hypertension
* coronary artery disease
* cerebral disease
* COPD/asthma
* oral/pharyngeal/laryngeal carcinoma
* loose teeth/poor dentition
* Macintosh laryngoscope >size 3 required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-02 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Forces generated during the intubation process using both laryngoscopes including peak and mean forces. | 5-15minutes

CONTACTS AND LOCATIONS:
Overall Officials: Richard Cooper, MD, Principal Investigator — Toronto General Hospital, University Health Network
Locations (2):
- Canada (2):
  - Toronto General Hospital, UHN, Toronto, Ontario
  - Toronto General Hospital, University Health Network, Toronto, Ontario